CLINICAL TRIAL: NCT04590807
Title: Posterior Spinal Fusion With Pedicle Screws vs. Anterior Vertebral Body Tethering in Adolescent Idiopathic Scoliosis (AIS): an International Multicenter Randomized Clinical Trial
Brief Title: Posterior Spinal Fusion With Pedicle Screws vs. Anterior Vertebral Body Tethering in Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Ilkka Helenius, MD, PhD, Professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETMK 15/1801/2020
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Spinal Diseases
MeSH Terms: conditions — Scoliosis; Spinal Diseases | interventions — Pedicle Screws

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior spinal fusion with pedicle screws (Active Comparator)
  Interventions: Device: Posterior spinal fusion with pedicle screws
- Anterior vertebral body tethering (Active Comparator)
  Interventions: Device: Anterior vertebral body tethering

INTERVENTIONS:
Device: Posterior spinal fusion with pedicle screws — Implanting pedicle screws and rods
  Arms: Posterior spinal fusion with pedicle screws
Device: Anterior vertebral body tethering — Vertebral screws and cable
  Arms: Anterior vertebral body tethering

SUMMARY:
Background- Adolescent idiopathic scoliosis is the most common indication for major surgery in adolescents. The current standard of care for adolescent idiopathic scoliosis (AIS) with a curve magnitude of over 40-50˚ in skeletally immature patients, is posterior spinal fusion with pedicle screws. Vertebral body tethering using screws connected by a tether in the anterior vertebral body, has the potential to initially correct the still flexible deformity, but most importantly modulate growth and ultimately result in scoliosis correction with a mobile spine. A high-quality comparative prospective study is missing to demonstrate the effectiveness and safety of vertebral body tethering compared to posterior spinal fusion.

Study Design- An international, randomized clinical trial on posterior spinal fusion with pedicle screws vs. Anterior vertebral body tethering in Adolescent Idiopathic Scoliosis (AIS)

Aims- To demonstrate non-inferiority of VBT compared to posterior fusion in terms of main curve correction of AIS at the 2 year follow up, to demonstrate comparable outcomes for SRS-22/24 at the 2 year follow up. Aim is also to compare complication and revision rates and to compare spinal mobility including flexion and side bending between the study groups.

Inclusion criteria- Lenke type I A,B or C, age 10-16 years, skeletally immature, Cobb angle 40-60˚, 50% flexibility on supine bending films, selective thoracic fusion feasible

Exclusion criteria- Any other than idiopathic scoliosis, less than 50% curve flexibility, skeletal maturity, patients who have evidence of neurological disorders, patients who have undergone intrathoracic surgery

Outcome parametres- Cobb angle correction of instrumented curve at 2 year follow up, total score of SRS questionnaire at 2 year follow up; secondary outcomes: Complication and revision rates, pulmonary function at 2-year follow-up, spinal mobility at 2-year follow-up

Ethical aspects- Each institution in each country is responsible for obtaining either institutional review board approval or approval from a national ethics committee as appropriate. An informed consent will be obtained from all children and their parents.

DETAILED DESCRIPTION:
Background- Adolescent idiopathic scoliosis is the most common indication for major surgery in adolescents (between 10 and 18 years of age). The current standard of care for adolescent idiopathic scoliosis (AIS) with a curve magnitude of over 40-50˚ in skeletally immature patients, is posterior spinal fusion with pedicle screws. The aim of spinal fusion is to prevent further curve progression but also to correct the spinal deformity and achieve a cosmetically pleasing result by reducing the rib hump and balancing the trunk and shoulders. While this procedure has been very successful, it has inherent downsides such as the decreased range of motion and loss of spinal mobility in addition to the inhibition of growth along the instrumentation. To prevent distal adding on (continued curve below instrumentation) due to continued anterior spinal growth, it is often necessary to fuse the spine into stable vertebra resulting into even longer spinal fusion levels in the lumbar spine (Sponseller et al. JPO 2016; Oksanen et al. SJS 2018). Spinal fusion increases loading of the remaining mobile segments (Parsch et al. JBJS Br 2001).

In a five-year follow-up study spinal fusion resulted into better health-related quality of life (HRQoL) as compared with untreated AIS (Helenius et al. JBJS 2019). However, the function domain of HRQoL was significantly less after spinal fusion as compared with healthy controls. In contrast, vertebral body tethering using screws connected by a tether in the anterior vertebral body, has the potential to initially correct the still flexible deformity, but most importantly modulate growth and ultimately result in scoliosis correction with a mobile spine.

There is currently a paucity of literature on the effectiveness of vertebral body tethering (VBT) with only retrospective case series published and reported in conference proceedings, and a comparative study is completely lacking. Initial complication rates with the implants for tethering have also sparked caution amongst surgeons and payers whether or not to adopt this technique despite its theoretical advantages. Thus, a high-quality comparative prospective study is missing to demonstrate the effectiveness and safety of vertebral body tethering compared to posterior spinal fusion. If this can be shown in a well-designed study, it is likely to result in a paradigm shift in the treatment of AIS similar to the impact earlier technical novelties and achievements had.

Randomised controlled trials are rare in paediatric orthopaedic research. It would be unprecedented that evidence from an RCT is driving a change in practice in scoliosis surgery.

Aims and hypothesis- To compare posterior fusion to VBT for the treatment of AIS. Aim is to demonstrate non-inferiority of VBT compared to posterior fusion in terms of main curve correction of AIS at the 2 year follow up, to demonstrate comparable outcomes for SRS-22/24 at the 2 year follow up. Aim is also to compare complication and revision rates and to compare spinal mobility including flexion and side bending between the study groups.

Inclusion criteria- The inclusion criteria would aim to restrict the study to paediatric patients with AIS and the following criteria: Lenke type I A,B or C, age 10-16 years, skeletally immature (Sanders classification between 2 and 5), Cobb angle 40-60˚, 50% flexibility on supine bending films, selective thoracic fusion feasible

Exclusion criteria- Any other than idiopathic scoliosis, less than 50% curve flexibility, skeletal maturity (Sanders >5), patients who have evidence of neurological disorders, patients who have undergone intrathoracic surgery Outcome parametres- Cobb angle correction of instrumented curve at 2 year follow up, total score of SRS questionnaire at 2 year follow up; secondary outcomes: Complication and revision rates, pulmonary function at 2-year follow-up, spinal mobility at 2-year follow-up

Interventions: AVBT from end to end vertebra. PSF levels using the Lenke criteria.

Ethical aspects- Each institution in each country is responsible for obtaining either institutional review board approval or approval from a national ethics committee as appropriate. An informed consent will be obtained from all children and their parents.

Time schedule and budget- The study will be started on beginning of 2021. Patient enrollment is expected to last to the end of 2023. There will be no extra costs as all information gathered will be part of normal surgical treatment of AIS. A part-time research nurse has been hired to take care of data collection into the database.

References:

1. Sponseller PD, Jain A, Newton PO et al. Posterior Spinal Fusion With Pedicle Screws in Patients With Idiopathic Scoliosis and Open Triradiate Cartilage: Does Deformity Progression Occur? J Pediatr Orthop 2016; 36:695-700.
2. Oksanen H, Lastikka M, Helenius L, et al. Posterior Spinal Fusion Extended to Stable Vertebra Provides Similar Outcome in Juvenile Idiopathic Scoliosis Patients Compared with Adolescents with Fusion to the Touched Vertebra. Scand J Surg 2019 Mar; 108(1):83-89.
3. Parsch et al. JBJS Br 2001
4. Helenius L, Diabakerli E, Grauers A, et al. Back Pain and Quality of Life after Surgical Treatment for Adolescent Idiopathic Scoliosis

ELIGIBILITY:
Inclusion Criteria:

* AIS Lenke type I A,B or C
* Age 10-16 years
* Skeletally immature (Sanders classification between 2 and 5)
* Cobb angle 40-60˚
* 50% flexibility on supine bending films.
* Selective thoracic fusion feasible

Exclusion Criteria:

* Any other than idiopathic scoliosis
* Less than 50% curve flexibility
* Skeletal maturity (Sanders >5)
* Patients who have evidence of neurological disorders
* Patients who have undergone intrathoracic surgery

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cobb angle correction of instrumented curve at 2 year follow up | 2 years follow-up
  Major Curve Cobb Angle (Cobb, 1948)
Total score of SRS-24 questionnaire at 2 year follow up | 2 years follow-up
  SRS-24 outcome questionnaire. Total score between 1 to 5

SECONDARY OUTCOMES:
Complication rate | 2 years follow-up
  deep surgical site infection, neurologic deficit
Revision rate | 2 years follow-up
  Any re-intervention
Pulmonary function at 2-year follow-up | 2 years follow-up
  FVC (% predicted)
Spinal mobility at 2-year follow-up | 2 years follow-up
  Trunk side bending (finger tip to knee joint, cm), forward bending (finger tip to floor distance, cm)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Newton PO, Kluck DG, Saito W, Yaszay B, Bartley CE, Bastrom TP. Anterior Spinal Growth Tethering for Skeletally Immature Patients with Scoliosis: A Retrospective Look Two to Four Years Postoperatively. J Bone Joint Surg Am. 2018 Oct 3;100(19):1691-1697. doi: 10.2106/JBJS.18.00287. PMID 30277999
- [Result] Wong HK, Ruiz JNM, Newton PO, Gabriel Liu KP. Non-Fusion Surgical Correction of Thoracic Idiopathic Scoliosis Using a Novel, Braided Vertebral Body Tethering Device: Minimum Follow-up of 4 Years. JB JS Open Access. 2019 Dec 12;4(4):e0026. doi: 10.2106/JBJS.OA.19.00026. eCollection 2019 Oct-Dec. PMID 32043058
- [Result] Newton PO, Bartley CE, Bastrom TP, Kluck DG, Saito W, Yaszay B. Anterior Spinal Growth Modulation in Skeletally Immature Patients with Idiopathic Scoliosis: A Comparison with Posterior Spinal Fusion at 2 to 5 Years Postoperatively. J Bone Joint Surg Am. 2020 May 6;102(9):769-777. doi: 10.2106/JBJS.19.01176. PMID 32379117